CLINICAL TRIAL: NCT03269708
Title: Improving Cardiac Secondary Prevention Through Personalized Biomarker Knowledge
Brief Title: Improving Cardiac Secondary Prevention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Geoffrey Pickering MD PhD, Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 109209
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Myocardial Infarction; Secondary Prevention
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants receive standard care in cardiac rehabilitation program
- Knowledge transfer group (Experimental): Participants receive standard care in cardiac rehabilitation program plus education regarding telomere length
  Interventions: Behavioral: Education regarding telomere length

INTERVENTIONS:
Behavioral: Education regarding telomere length — Teaching concepts of cellular aging and telomere length
  Arms: Knowledge transfer group

SUMMARY:
The purpose of this study is to determine whether providing individuals with personalized information on cellular aging, including telomere length, will stimulate them to adhere to cardiac prevention strategies and improve exercise capacity.

DETAILED DESCRIPTION:
Individuals who have sustained a heart attack are at considerable risk for future cardiac events. A cardiac rehabilitation and exercise program can reduce this risk but it remains a challenge to adopt optimum lifestyle changes. We will determine whether providing individuals with information on leukocyte telomere length, will motivate them to improve their exercise performance. We will test whether professionally conveying this information will stimulate an individual to adhere to proven cardiac prevention strategies, looking at the extent to which one's exercise capacity improves over time.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who have sustained a myocardial infarction and entered the cardiac rehabilitation program

Exclusion Criteria:

1. Individuals with genetic mutations that affect telomere length
2. Individuals who may not have the mental capacity to understanding the ramifications of risk biomarkers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity based on cardiopulmonary exercise testing | after 6-month cardiac rehabilitation program
  Online VO2 maximum

SECONDARY OUTCOMES:
Adherence to supervised exercise sessions | 6 months
  Proportion of prescribed supervised on-site exercise sessions attended
Activity assessment | 6 months
  Garmin recording

CONTACTS AND LOCATIONS:
Overall Officials: J. Geoffrey Pickering, MD PhD, Principal Investigator — Western Faculty
Locations (1):
- London Health Sciences Centre, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No